CLINICAL TRIAL: NCT00212134
Title: Infant Aphakia Treatment Study (IATS)
Acronym: IATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Alcon Research (Industry); Bausch & Lomb Incorporated (Industry); BSN-JOBST Inc. (Industry); Eye Care and Cure (Industry)
Responsible Party: Principal Investigator, Scott Reed Lambert, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024837; U10EY013272 (NIH); EY013287 (Other Grant/Funding Number: Emory); EY013272 (Other Grant/Funding Number: Emory); NEI-108 (Other: Other)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Congenital Cataract
Keywords: cataract surgery; intraocular lens; contact lens; infants; aphakia
MeSH Terms: conditions — Aphakia | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: Phase 3 is 10.5-year follow-up study since Phase 1. There is no intervention.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aphakic contact lens (Active Comparator): Contact lens correction of aphakia
  INTERVENTION: use of an external contact lens (CL) to correct the large hyperopic refractive error produced by surgically extracting the natural cataractous lens. As the eye grows, the refractive error changes and the power of the CL can be changed accordingly.
  Interventions: Device: Contact lens correction of aphakia
- aphakic intraocular lens (Experimental): Intraocular lens implantation
  INTERVENTION: At the time of surgery to remove the cataractous natural lens, an intraocular lens was implanted to correct the large hyperopic refractive error induced by the cataract surgery.
  Interventions: Device: Intraocular lens implantation

INTERVENTIONS:
Device: Contact lens correction of aphakia — optical correction of infant surgical aphakia with Contact lens
  Other Names: Silsoft aphakic contact lens; rigid gas permeable contact lens
  Arms: aphakic contact lens
Device: Intraocular lens implantation — optical correction of surgical aphakia with intraocular lens
  Other Names: Alcon SA60AT; Alcon MA60AC
  Arms: aphakic intraocular lens

SUMMARY:
The primary purpose is to determine whether infants with a unilateral congenital cataract are more likely to develop better vision following cataract extraction surgery if they undergo primary implantation of an intraocular lens or if they are treated primarily with a contact lens. In addition, the study will compare the occurrence of postoperative complications and the degree of parental stress between the two treatments.

DETAILED DESCRIPTION:
Intraocular lenses are now a commonly accepted treatment for cataracts in older children and are used increasingly in younger children and infants. Intraocular lenses are superior to contact lenses in that they more closely replicate the optics of the crystalline lens, do not require daily ongoing care, and ensure at least a partial optical correction at all times. The simplicity and improved visual outcome of an intraocular lens correction may make caring for a child with a unilateral congenital cataract less stressful for parents. However, contact lenses remain the accepted treatment for children under 1 year of age due to concerns about the long-term safety of intraocular lenses and the potential for a large myopic shift developing in these eyes as they grow. Contact lenses provide excellent visual results in infants treated for bilateral congenital cataracts; however, two-thirds of infants treated with contact lenses for unilateral congenital cataracts remain legally blind in their aphakic eye. These poor visual outcomes are usually ascribed to competition from the sound eye and poor compliance with patching and contact lens wear regimens. Data from our pilot study and the literature suggest that superior visual results can be obtained if an intraocular lens is used to correct unilateral aphakia during infancy, but these eyes will experience more complications. Intraocular lenses will be increasingly implanted in infants regardless of whether or not we perform this trial. By performing this clinical trial, we can determine if the higher rate of complications with intraocular lenses is offset by improved visual outcome and decreased parenting stress.

The Infant Aphakia Treatment Study (IATS) is a multi-center randomized clinical trial comparing intraocular lens and contact lens correction for monocular aphakia. Infants will be enrolled over a 4 year period. Infants 28 to 210 days of age with a visually significant cataract in one eye are eligible. Cataract surgery will be performed in a standardized fashion by a surgeon who has been certified for the study. Surgery consists of a lensectomy, posterior capsulotomy, and anterior vitrectomy. Infants will be randomized at the time of surgery to one of two treatment groups. Infants randomized to the intraocular lens group will have an intraocular lens implanted into the capsular bag. Spectacles will subsequently be used to correct the residual refractive errors. Infants randomized to the contact lens group will be fitted with a contact lens immediately after surgery. Both groups will receive the same patching therapy and follow-up. All children will be examined by Investigators at fixed intervals using standard protocols with the major endpoint assessed at age 12 months by a Traveling Vision Examiner.

We are currently in a continuation of this project (beyond 5 years) in order to assess which of these patients have glaucoma or glaucoma suspect at age 10.5 years. Our goal is to understand which type of initial optical correction, an IOL or a CL, results in the best long-term visual outcome following unilateral congenital cataract surgery during infancy. Our central hypothesis is that primary IOL implantation will result in a better visual outcome. The rationale for this proposal is that final visual acuity cannot be determined by 5 years of age and the recommendation for early treatment can only be substantiated by adequate long-term assessment in this unique cohort. We chose a follow-up to age 10.5 years because it will provide a more accurate assessment of visual acuity and will allow us to diagnosis most cases of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Visually significant unilateral congenital cataract (central opacity equal to or greater than 3 mm in size).
* Cataract surgery performed when the patient is 28 to 210 days of age and at least 41 post-conceptional weeks.

Exclusion Criteria:

* The cataract is known to be acquired from trauma or as a side-effect of a treatment administered postnatally such as radiation or medical therapy.
* A corneal diameter less than 9 mm measured in the horizontal meridian using calipers.
* An intraocular pressure of 25 mm Hg or greater in the affected eye measured with a Perkins tonometer, tonopen, or pneumatonometer.
* Persistent fetal vasculature (PFV) causing stretching of the ciliary processes or a tractional retinal detachment.
* Active uveitis or signs suggestive of a previous episode of uveitis such as posterior synechiae or keratic precipitates.
* The child is the product of a pre-term pregnancy (<36 gestational weeks). Screening for prematurity will be based on the clinician's best assessment of gestational age. If a physician is uncertain regarding the gestational age, review of medical records or contact with the pediatrician and/or obstetrician should be used to confirm gestational age at delivery. Unless a clinician is uncertain as to whether a child was born at less than 36 weeks or not, confirmation of gestational age via medical record review may be delayed until after enrollment.
* Retinal disease that may limit the visual potential of the eye such as retinopathy of prematurity.
* Previous intraocular surgery.
* Optic nerve disease that may limit the visual potential of the eye such as optic nerve hypoplasia.
* The fellow eye has ocular disease that might reduce its visual potential.
* The child has a medical condition known to limit the ability to obtain visual acuity at 12 months or 4 years of age.
* Refusal by the Parent/Legal Guardian to sign an informed consent or to be randomized to one of the two treatment groups.
* Follow-up of the child is not feasible because the child would not be able to return for regular follow-up examinations and the outcome assessments (e.g. transportation difficulties, relocation, etc.).

Ages: 28 Days to 210 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lambert, MD, Study Chair — Stanford University
Locations (13):
- United States (13):
  - Stanford University, Palo Alto, California
  - Miami Children's Hospital, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Indiana University Medical Center, Indianapolis, Indiana
  - Harvard University, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University Eye Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Pediatric Ophthalmology, P.A., Dallas, Texas
  - Baylor University, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bothun ED, Lynn MJ, Lambert SR. Author reply: To PMID 23419803. Ophthalmology. 2014 Oct;121(10):e53. doi: 10.1016/j.ophtha.2014.05.011. Epub 2014 Jun 6. No abstract available. PMID 24909820
- [Result] Traboulsi EI, Vanderveen D, Morrison D, Drews-Botsch CD, Lambert SR; Infant Aphakia Treatment Study Group. Associated systemic and ocular disorders in patients with congenital unilateral cataracts: the Infant Aphakia Treatment Study experience. Eye (Lond). 2016 Sep;30(9):1170-4. doi: 10.1038/eye.2016.124. Epub 2016 Jun 17. PMID 27315350
- [Result] Drews-Botsch C, Celano M, Cotsonis G, Hartmann EE, Lambert SR; Infant Aphakia Treatment Study Group. Association Between Occlusion Therapy and Optotype Visual Acuity in Children Using Data From the Infant Aphakia Treatment Study: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2016 Aug 1;134(8):863-9. doi: 10.1001/jamaophthalmol.2016.1365. PMID 27228110
- [Result] Lambert SR, Plager DA, Lynn MJ, Wilson ME. Visual outcome following the reduction or cessation of patching therapy after early unilateral cataract surgery. Arch Ophthalmol. 2008 Aug;126(8):1071-4. doi: 10.1001/archopht.126.8.1071. PMID 18695101
- [Result] Infant Aphakia Treatment Study Group; Lambert SR, Buckley EG, Drews-Botsch C, DuBois L, Hartmann E, Lynn MJ, Plager DA, Wilson ME. The infant aphakia treatment study: design and clinical measures at enrollment. Arch Ophthalmol. 2010 Jan;128(1):21-7. doi: 10.1001/archophthalmol.2009.350. PMID 20065212
- [Result] Infant Aphakia Treatment Study Group; Lambert SR, Buckley EG, Drews-Botsch C, DuBois L, Hartmann EE, Lynn MJ, Plager DA, Wilson ME. A randomized clinical trial comparing contact lens with intraocular lens correction of monocular aphakia during infancy: grating acuity and adverse events at age 1 year. Arch Ophthalmol. 2010 Jul;128(7):810-8. doi: 10.1001/archophthalmol.2010.101. Epub 2010 May 10. PMID 20457949
- [Result] Plager DA, Lynn MJ, Buckley EG, Wilson ME, Lambert SR; Infant Aphakia Treatment Study Group. Complications, adverse events, and additional intraocular surgery 1 year after cataract surgery in the infant Aphakia Treatment Study. Ophthalmology. 2011 Dec;118(12):2330-4. doi: 10.1016/j.ophtha.2011.06.017. Epub 2011 Sep 16. PMID 21925737
- [Result] Morrison DG, Wilson ME, Trivedi RH, Lambert SR, Lynn MJ; Infant Aphakia Treatment Study Group. Infant Aphakia Treatment Study: effects of persistent fetal vasculature on outcome at 1 year of age. J AAPOS. 2011 Oct;15(5):427-31. doi: 10.1016/j.jaapos.2011.06.004. PMID 22108353
- [Result] Wilson ME, Trivedi RH, Morrison DG, Lambert SR, Buckley EG, Plager DA, Lynn MJ; Infant Aphakia Treatment Study Group. The Infant Aphakia Treatment Study: evaluation of cataract morphology in eyes with monocular cataracts. J AAPOS. 2011 Oct;15(5):421-6. doi: 10.1016/j.jaapos.2011.05.016. PMID 22108352
- [Result] Drews-Botsch CD, Hartmann EE, Celano M; Infant Aphakia Treatment Study Group. Predictors of adherence to occlusion therapy 3 months after cataract extraction in the Infant Aphakia Treatment Study. J AAPOS. 2012 Apr;16(2):150-5. doi: 10.1016/j.jaapos.2011.12.149. PMID 22525171
- [Result] Beck AD, Freedman SF, Lynn MJ, Bothun E, Neely DE, Lambert SR; Infant Aphakia Treatment Study Group. Glaucoma-related adverse events in the Infant Aphakia Treatment Study: 1-year results. Arch Ophthalmol. 2012 Mar;130(3):300-5. doi: 10.1001/archophthalmol.2011.347. Epub 2011 Nov 14. PMID 22084157
- [Result] VanderVeen DK, Nizam A, Lynn MJ, Bothun ED, McClatchey SK, Weakley DR, DuBois LG, Lambert SR; Infant Aphakia Treatment Study Group. Predictability of intraocular lens calculation and early refractive status: the Infant Aphakia Treatment Study. Arch Ophthalmol. 2012 Mar;130(3):293-9. doi: 10.1001/archophthalmol.2011.358. PMID 22411658
- [Result] Russell B, Ward MA, Lynn M, Dubois L, Lambert SR; Infant Aphakia Treatment Study Group. The infant aphakia treatment study contact lens experience: one-year outcomes. Eye Contact Lens. 2012 Jul;38(4):234-9. doi: 10.1097/ICL.0b013e3182562dc0. PMID 22669008
- [Result] Lambert SR, Purohit A, Superak HM, Lynn MJ, Beck AD. Long-term risk of glaucoma after congenital cataract surgery. Am J Ophthalmol. 2013 Aug;156(2):355-361.e2. doi: 10.1016/j.ajo.2013.03.013. Epub 2013 Apr 30. PMID 23639132
- [Result] Carrigan AK, DuBois LG, Becker ER, Lambert SR; Infant Aphakia Treatment Study Group. Cost of intraocular lens versus contact lens treatment after unilateral congenital cataract surgery: retrospective analysis at age 1 year. Ophthalmology. 2013 Jan;120(1):14-9. doi: 10.1016/j.ophtha.2012.07.049. Epub 2012 Oct 6. PMID 23047003
- [Result] Trivedi RH, Lambert SR, Lynn MJ, Wilson ME; Infant Aphakia Treatment Study Group. The role of preoperative biometry in selecting initial contact lens power in the Infant Aphakia Treatment Study. J AAPOS. 2014 Jun;18(3):251-4. doi: 10.1016/j.jaapos.2014.01.012. PMID 24924278
- [Result] Vanderveen DK, Trivedi RH, Nizam A, Lynn MJ, Lambert SR; Infant Aphakia Treatment Study Group. Predictability of intraocular lens power calculation formulae in infantile eyes with unilateral congenital cataract: results from the Infant Aphakia Treatment Study. Am J Ophthalmol. 2013 Dec;156(6):1252-1260.e2. doi: 10.1016/j.ajo.2013.07.014. Epub 2013 Sep 4. PMID 24011524
- [Result] Hartmann EE, Stout AU, Lynn MJ, Yen KG, Kruger SJ, Lambert SR; Infant Aphakia Treatment Study Group; Infant Aphakia Treatment Study Group. Stereopsis results at 4.5 years of age in the infant aphakia treatment study. Am J Ophthalmol. 2015 Jan;159(1):64-70.e1-2. doi: 10.1016/j.ajo.2014.09.028. Epub 2014 Sep 28. PMID 25261241
- [Result] Infant Aphakia Treatment Study Group; Lambert SR, Lynn MJ, Hartmann EE, DuBois L, Drews-Botsch C, Freedman SF, Plager DA, Buckley EG, Wilson ME. Comparison of contact lens and intraocular lens correction of monocular aphakia during infancy: a randomized clinical trial of HOTV optotype acuity at age 4.5 years and clinical findings at age 5 years. JAMA Ophthalmol. 2014 Jun;132(6):676-82. doi: 10.1001/jamaophthalmol.2014.531. PMID 24604348
- [Result] Kruger SJ, DuBois L, Becker ER, Morrison D, Wilson L, Wilson ME Jr, Lambert SR; Infant Aphakia Treatment Study Group. Cost of intraocular lens versus contact lens treatment after unilateral congenital cataract surgery in the infant aphakia treatment study at age 5 years. Ophthalmology. 2015 Feb;122(2):288-92. doi: 10.1016/j.ophtha.2014.08.037. Epub 2014 Oct 29. PMID 25439604
- [Result] Wall PB, Lee JA, Lynn MJ, Lambert SR, Traboulsi EI; Infant Aphakia Treatment Study Group. The effects of surgical factors on postoperative astigmatism in patients enrolled in the Infant Aphakia Treatment Study (IATS). J AAPOS. 2014 Oct;18(5):441-5. doi: 10.1016/j.jaapos.2014.06.016. Epub 2014 Sep 27. PMID 25266831
- [Result] Bothun ED, Cleveland J, Lynn MJ, Christiansen SP, Vanderveen DK, Neely DE, Kruger SJ, Lambert SR; Infant Aphakic Treatment Study. One-year strabismus outcomes in the Infant Aphakia Treatment Study. Ophthalmology. 2013 Jun;120(6):1227-31. doi: 10.1016/j.ophtha.2012.11.039. Epub 2013 Feb 16. PMID 23419803
- [Result] Freedman SF, Lynn MJ, Beck AD, Bothun ED, Orge FH, Lambert SR; Infant Aphakia Treatment Study Group. Glaucoma-Related Adverse Events in the First 5 Years After Unilateral Cataract Removal in the Infant Aphakia Treatment Study. JAMA Ophthalmol. 2015 Aug;133(8):907-14. doi: 10.1001/jamaophthalmol.2015.1329. PMID 25996491
- [Result] Plager DA, Lynn MJ, Buckley EG, Wilson ME, Lambert SR; Infant Aphakia Treatment Study Group. Complications in the first 5 years following cataract surgery in infants with and without intraocular lens implantation in the Infant Aphakia Treatment Study. Am J Ophthalmol. 2014 Nov;158(5):892-8. doi: 10.1016/j.ajo.2014.07.031. Epub 2014 Jul 29. PMID 25077835
- [Result] Morrison DG, Lynn MJ, Freedman SF, Orge FH, Lambert SR; Infant Aphakia Treatment Study Group. Corneal Changes in Children after Unilateral Cataract Surgery in the Infant Aphakia Treatment Study. Ophthalmology. 2015 Nov;122(11):2186-92. doi: 10.1016/j.ophtha.2015.07.011. Epub 2015 Aug 11. PMID 26271843
- [Result] VanderVeen DK, Trivedi RH, Nizam A, Lynn MJ, Lambert SR. Reply: To PMID 24011524. Am J Ophthalmol. 2014 Jun;157(6):1332-3. doi: 10.1016/j.ajo.2014.02.053. No abstract available. PMID 24881851
- [Result] Kumar P, Lambert SR. Evaluating the evidence for and against the use of IOLs in infants and young children. Expert Rev Med Devices. 2016;13(4):381-9. doi: 10.1586/17434440.2016.1153967. Epub 2016 Feb 29. PMID 26878234
- [Result] Bothun ED, Lynn MJ, Christiansen SP, Neely DE, Vanderveen DK, Kruger SJ, Lambert SR; Infant Aphakia Treatment Study. Sensorimotor outcomes by age 5 years after monocular cataract surgery in the Infant Aphakia Treatment Study (IATS). J AAPOS. 2016 Feb;20(1):49-53. doi: 10.1016/j.jaapos.2015.11.002. PMID 26917072
- [Result] Celano M, Hartmann EE, DuBois LG, Drews-Botsch C; Infant Aphakia Treatment Study Group. Motor skills of children with unilateral visual impairment in the Infant Aphakia Treatment Study. Dev Med Child Neurol. 2016 Feb;58(2):154-9. doi: 10.1111/dmcn.12832. Epub 2015 Jun 17. PMID 26084944
- [Result] Lambert SR, Plager DA, Buckley EG, Wilson ME, DuBois L, Drews-Botsch CD, Hartmann EE, Lynn MJ; Infant Aphakia Treatment Study Group. The Infant Aphakia Treatment Study: further on intra- and postoperative complications in the intraocular lens group. J AAPOS. 2015 Apr;19(2):101-3. doi: 10.1016/j.jaapos.2015.01.012. No abstract available. PMID 25892038
- [Result] Lambert SR, Lynn MJ, Hartmann EE; Infant Aphakia Treatment Study Group. In reply. JAMA Ophthalmol. 2014 Dec;132(12):1492-3. doi: 10.1001/jamaophthalmol.2014.3542. No abstract available. PMID 25256439
- [Result] Celano M, Hartmann EE, Drews-Botsch CD; Infant Aphakia Treatment Study Group. Parenting stress in the infant aphakia treatment study. J Pediatr Psychol. 2013 Jun;38(5):484-93. doi: 10.1093/jpepsy/jst009. Epub 2013 Mar 9. PMID 23475835
- [Result] Lenhart PD, Courtright P, Wilson ME, Lewallen S, Taylor DS, Ventura MC, Bowman R, Woodward L, Ditta LC, Kruger S, Haddad D, El Shakankiri N, Rai SK, Bailey T, Lambert SR. Global challenges in the management of congenital cataract: proceedings of the 4th International Congenital Cataract Symposium held on March 7, 2014, New York, New York. J AAPOS. 2015 Apr;19(2):e1-8. doi: 10.1016/j.jaapos.2015.01.013. PMID 25892047
- [Result] Nguyen M, Shainberg M, Beck AD, Lambert SR. Structural changes of the anterior chamber following cataract surgery during infancy. J Cataract Refract Surg. 2015 Aug;41(8):1784-6. doi: 10.1016/j.jcrs.2015.07.001. No abstract available. PMID 26432141
- [Result] Russell B, DuBois L, Lynn M, Ward MA, Lambert SR; Infant Aphakia Treatment Study Group. The Infant Aphakia Treatment Study Contact Lens Experience to Age 5 Years. Eye Contact Lens. 2017 Nov;43(6):352-357. doi: 10.1097/ICL.0000000000000291. PMID 27466719
- [Result] Lambert SR. The timing of surgery for congenital cataracts: Minimizing the risk of glaucoma following cataract surgery while optimizing the visual outcome. J AAPOS. 2016 Jun;20(3):191-2. doi: 10.1016/j.jaapos.2016.04.003. Epub 2016 May 11. No abstract available. PMID 27180288
- [Result] Celano M, Cotsonis GA, Hartmann EE, Drews-Botsch C; Infant Aphakia Treatment Study Group. Behaviors of children with unilateral vision impairment in the Infant Aphakia Treatment Study. J AAPOS. 2016 Aug;20(4):320-5. doi: 10.1016/j.jaapos.2016.04.008. Epub 2016 Jul 14. PMID 27424046
- [Result] Drews-Botsch C, Cotsonis G, Celano M, Lambert SR. Assessment of Adherence to Visual Correction and Occlusion Therapy in the Infant Aphakia Treatment Study. Contemp Clin Trials Commun. 2016 Aug 15;3:158-166. doi: 10.1016/j.conctc.2016.05.009. Epub 2016 May 30. PMID 27981259
- [Result] Lambert SR, DuBois L, Cotsonis G, Hartmann EE, Drews-Botsch C. Factors associated with stereopsis and a good visual acuity outcome among children in the Infant Aphakia Treatment Study. Eye (Lond). 2016 Sep;30(9):1221-8. doi: 10.1038/eye.2016.164. Epub 2016 Jul 29. PMID 27472216
- [Result] Bothun ED, Lynn MJ, Christiansen SP, Kruger SJ, Vanderveen DK, Neely DE, Lambert SR; Infant Aphakic Treatment Study. Strabismus surgery outcomes in the Infant Aphakia Treatment Study (IATS) at age 5 years. J AAPOS. 2016 Dec;20(6):501-505. doi: 10.1016/j.jaapos.2016.09.014. Epub 2016 Nov 2. PMID 27815186
- [Result] Lambert SR, Cotsonis G, DuBois L, Wilson ME, Plager DA, Buckley EG, McClatchey SK; Infant Aphakia Treatment Study Group. Comparison of the rate of refractive growth in aphakic eyes versus pseudophakic eyes in the Infant Aphakia Treatment Study. J Cataract Refract Surg. 2016 Dec;42(12):1768-1773. doi: 10.1016/j.jcrs.2016.09.021. PMID 28007108
- [Result] Cooke DL. Predictability of intraocular lens power calculation formulae in infantile eyes with unilateral congenital cataract: results from the infant aphakia treatment study. Am J Ophthalmol. 2014 Jun;157(6):1332. doi: 10.1016/j.ajo.2014.02.051. No abstract available. PMID 24881852
- [Result] Drews-Botsch CD, Celano M, Kruger S, Hartmann EE; Infant Aphakia Treatment Study. Adherence to occlusion therapy in the first six months of follow-up and visual acuity among participants in the Infant Aphakia Treatment Study (IATS). Invest Ophthalmol Vis Sci. 2012 Jun 5;53(7):3368-75. doi: 10.1167/iovs.11-8457. PMID 22491410
- [Result] Felius J, Busettini C, Lynn MJ, Hartmann EE, Lambert SR; Infant Aphakia Treatment Study Group. Nystagmus and related fixation instabilities following extraction of unilateral infantile cataract in the Infant Aphakia Treatment Study (IATS). Invest Ophthalmol Vis Sci. 2014 Aug 5;55(8):5332-7. doi: 10.1167/iovs.14-14710. PMID 25097243
- [Result] Lambert SR, Lynn MJ, DuBois LG, Cotsonis GA, Hartmann EE, Wilson ME; Infant Aphakia Treatment Study Groups. Axial elongation following cataract surgery during the first year of life in the infant Aphakia Treatment Study. Invest Ophthalmol Vis Sci. 2012 Nov 7;53(12):7539-45. doi: 10.1167/iovs.12-10285. PMID 23074203
- [Result] Wilson ME, Trivedi RH, Weakley DR Jr, Cotsonis GA, Lambert SR; Infant Aphakia Treatment Study Group. Globe Axial Length Growth at Age 5 Years in the Infant Aphakia Treatment Study. Ophthalmology. 2017 May;124(5):730-733. doi: 10.1016/j.ophtha.2017.01.010. Epub 2017 Feb 10. PMID 28196730
- [Result] Weakley DR Jr, Lynn MJ, Dubois L, Cotsonis G, Wilson ME, Buckley EG, Plager DA, Lambert SR; Infant Aphakia Treatment Study Group. Myopic Shift 5 Years after Intraocular Lens Implantation in the Infant Aphakia Treatment Study. Ophthalmology. 2017 Jun;124(6):822-827. doi: 10.1016/j.ophtha.2016.12.040. Epub 2017 Feb 16. PMID 28215452
- [Result] Plager DA, Lynn MJ, Lambert SR, Buckley EG, Wilson ME; Infant Aphakia Treatment Study Group. Reply: To PMID 25077835. Am J Ophthalmol. 2014 Dec;158(6):1361-2. doi: 10.1016/j.ajo.2014.09.019. Epub 2014 Nov 18. No abstract available. PMID 25457713
- [Result] Weakley D, Cotsonis G, Wilson ME, Plager DA, Buckley EG, Lambert SR; Infant Aphakia Treatment Study Group. Anisometropia at Age 5 Years After Unilateral Intraocular Lens Implantation During Infancy in the Infant Aphakia Treatment Study. Am J Ophthalmol. 2017 Aug;180:1-7. doi: 10.1016/j.ajo.2017.05.008. Epub 2017 May 17. PMID 28526552
- [Result] Traboulsi EI, Freedman SF, Wilson ME Jr, Lambert SR; Infant Aphakia Treatment Study Group. Cataract morphology and risk for glaucoma after cataract surgery in infants with unilateral congenital cataract. J Cataract Refract Surg. 2017 Dec;43(12):1611-1612. doi: 10.1016/j.jcrs.2017.10.032. No abstract available. PMID 29335108
- [Result] Koo EB, VanderVeen DK, Lambert SR. Global Practice Patterns in the Management of Infantile Cataracts. Eye Contact Lens. 2018 Nov;44 Suppl 2(Suppl 2):S292-S296. doi: 10.1097/ICL.0000000000000461. PMID 29369235
- [Result] Cromelin CH, Drews-Botsch C, Russell B, Lambert SR; Infant Aphakia Treatment Study Group. Association of Contact Lens Adherence With Visual Outcome in the Infant Aphakia Treatment Study: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2018 Mar 1;136(3):279-285. doi: 10.1001/jamaophthalmol.2017.6691. PMID 29423513
- [Result] Weakley DR Jr, Lynn MJ, Dubois L, Cotsonis G, Wilson ME, Buckley EG, Plager DA, Lambert SR; Infant Aphakia Treatment Study Group. Reply. Ophthalmology. 2018 Oct;125(10):e69-e70. doi: 10.1016/j.ophtha.2018.03.058. No abstract available. PMID 30243340
- [Result] Hartmann EE, Drews-Botsch C, DuBois LG, Cotsonis G, Lambert SR; Infant Aphakia Treatment Study Group. Correlation of monocular grating acuity at age 12 months with recognition acuity at age 4.5 years: findings from the Infant Aphakia Treatment Study. J AAPOS. 2018 Aug;22(4):299-303.e2. doi: 10.1016/j.jaapos.2018.03.011. Epub 2018 Jul 20. PMID 30031874
- [Result] Lambert SR, DuBois L, Cotsonis G, Hartmann EE, Drews-Botsch C; Infant Aphakia Treatment Study Group. Spectacle Adherence Among Four-Year-Old Children in the Infant Aphakia Treatment Study. Am J Ophthalmol. 2019 Apr;200:26-33. doi: 10.1016/j.ajo.2018.12.017. Epub 2019 Jan 8. PMID 30633891
- [Result] Drews-Botsch C, Celano M, Cotsonis G, DuBois L, Lambert SR; Infant Aphakia Treatment Study Group. Parenting Stress and Adherence to Occlusion Therapy in the Infant Aphakia Treatment Study: A Secondary Analysis of a Randomized Clinical Trial. Transl Vis Sci Technol. 2019 Jan 2;8(1):3. doi: 10.1167/tvst.8.1.3. eCollection 2019 Jan. PMID 30627478
- [Result] Lambert SR, Bothun ED, Plager DA. Five-Year Postoperative Outcomes of Bilateral Aphakia and Pseudophakia in Children up to 2 Years of Age: A Randomized Clinical Trial. Am J Ophthalmol. 2019 Mar;199:263-264. doi: 10.1016/j.ajo.2018.09.042. Epub 2018 Dec 19. No abstract available. PMID 30579617
- [Result] Kruger SJ, Vanderveen DK, Freedman SF, Bothun E, Drews-Botsch CD, Lambert SR; Infant Aphakia Study Group. Third-Party Coverage for Aphakic Contact Lenses for Children. Transl Vis Sci Technol. 2019 Jun 14;8(3):41. doi: 10.1167/tvst.8.3.41. eCollection 2019 May. No abstract available. PMID 31231593
- [Result] Lambert SR, Cotsonis G, DuBois L, Nizam Ms A, Kruger SJ, Hartmann EE, Weakley DR Jr, Drews-Botsch C; Infant Aphakia Treatment Study Group. Long-term Effect of Intraocular Lens vs Contact Lens Correction on Visual Acuity After Cataract Surgery During Infancy: A Randomized Clinical Trial. JAMA Ophthalmol. 2020 Apr 1;138(4):365-372. doi: 10.1001/jamaophthalmol.2020.0006. PMID 32077909
- [Result] Lambert SR, Nizam A, DuBois L, Cotsonis G, Weakley DR Jr, Wilson ME; Infant Aphakia Treatment Study Group. The Myopic Shift in Aphakic Eyes in the Infant Aphakia Treatment Study After 10 Years of Follow-up. Eye Contact Lens. 2021 Feb 1;47(2):108-112. doi: 10.1097/ICL.0000000000000718. PMID 32568929
- [Result] Plager DA, Bothun ED, Freedman SF, Wilson ME, Lambert SR. Complications at 10 Years of Follow-up in the Infant Aphakia Treatment Study. Ophthalmology. 2020 Nov;127(11):1581-1583. doi: 10.1016/j.ophtha.2020.04.046. Epub 2020 May 11. No abstract available. PMID 32437863
- [Result] Traboulsi EI, Drews-Botsch CD, Christiansen SP, Stout AU, Hartmann EE, Lambert SR; IATS Investigator Group. Rate of ocular trauma in children operated on for unilateral cataract in infancy-data from the Infant Aphakia Treatment Study. J AAPOS. 2020 Oct;24(5):301-303. doi: 10.1016/j.jaapos.2020.06.005. Epub 2020 Aug 31. PMID 32882364
- [Result] VanderVeen DK, Drews-Botsch CD, Nizam A, Bothun ED, Wilson LB, Wilson ME, Lambert SR; Infant Aphakia Treatment Study. Outcomes of secondary intraocular lens implantation in the Infant Aphakia Treatment Study. J Cataract Refract Surg. 2021 Feb 1;47(2):172-177. doi: 10.1097/j.jcrs.0000000000000412. PMID 32925650
- [Result] McClatchey SK, McClatchey TS, Cotsonis G, Nizam A, Lambert SR; Infant Aphakia Treatment Study Group. Refractive growth variability in the Infant Aphakia Treatment Study. J Cataract Refract Surg. 2021 Apr 1;47(4):512-515. doi: 10.1097/j.jcrs.0000000000000482. PMID 33181631
- [Result] Freedman SF, Beck AD, Nizam A, Vanderveen DK, Plager DA, Morrison DG, Drews-Botsch CD, Lambert SR; Infant Aphakia Treatment Study Group. Glaucoma-Related Adverse Events at 10 Years in the Infant Aphakia Treatment Study: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2021 Feb 1;139(2):165-173. doi: 10.1001/jamaophthalmol.2020.5664. PMID 33331850
- [Result] Weakley DR Jr, Nizam A, VanderVeen DK, Wilson ME, Kruger S, Lambert SR; Infant Aphakia Treatment Study Group. Myopic Shift at 10-Year Follow-up in the Infant Aphakia Treatment Study. Ophthalmology. 2022 Sep;129(9):1064-1065. doi: 10.1016/j.ophtha.2022.04.004. Epub 2022 Apr 8. PMID 35398306
- [Result] Oke I, VanderVeen DK, McClatchey TS, Lambert SR, McClatchey SK; Infant Aphakia Treatment Study Group. The accuracy of intraocular lens calculation varies by age in the Infant Aphakia Treatment Study. J AAPOS. 2022 Jun;26(3):143-145. doi: 10.1016/j.jaapos.2022.02.004. Epub 2022 May 6. PMID 35534321
- [Result] Drews-Botsch C, Cotsonis G, Celano M, Hartmann EE, Zaidi J, Lambert SR. Patching in Children With Unilateral Congenital Cataract and Child Functioning and Parenting Stress. JAMA Ophthalmol. 2024 Jun 1;142(6):503-510. doi: 10.1001/jamaophthalmol.2024.0800. PMID 38635258
- [Derived] Wong C, Das U, Forbes H, Kolosky T, Cho E, Mansoor S, Chase S, Kore M, Menon R, Levin MR, Magder L, Drews-Botsch C, Lambert SR, Alexander JL. Predicting 10 Year Glaucoma Using Anterior Segment Biometry for Infants with Unilateral Congenital Cataract. Am J Ophthalmol. 2025 Dec 17;283:207-213. doi: 10.1016/j.ajo.2025.12.010. Online ahead of print. PMID 41419074
- [Derived] Hartmann EE, Drews-Botsch C, DuBois L, Lambert SR; Infant Aphakia Treatment Study Group. Stereopsis in the Infant Aphakia Treatment Study: outcome at 10(1/2) years. Eye (Lond). 2025 May;39(7):1426-1427. doi: 10.1038/s41433-025-03731-3. Epub 2025 Mar 8. PMID 40057655
- [Derived] Bothun ED, Shainberg MJ, Christiansen SP, Vanderveen DK, Neely DE, Kruger SJ, Cotsonis G, Lambert SR; Infant Aphakic Treatment Study. Long-term strabismus outcomes after unilateral infantile cataract surgery in the Infant Aphakia Treatment Study. J AAPOS. 2022 Aug;26(4):174.e1-174.e4. doi: 10.1016/j.jaapos.2022.05.003. Epub 2022 Jul 14. PMID 35843488
- [Derived] Hartmann EE, Lynn MJ, Lambert SR; Infant Aphakia Treatment Study Group. Baseline characteristics of the infant aphakia treatment study population: predicting recognition acuity at 4.5 years of age. Invest Ophthalmol Vis Sci. 2014 Dec 11;56(1):388-95. doi: 10.1167/iovs.14-15464. PMID 25503455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment 12/23/04 to 01/16/09 at 12 medical clinics.
Pre-assignment Details: Final eligibility determined at pre-operative ocular examination under anesthesia.
Groups:
- Aphakic Contact Lens: optical correction of infant aphakia with aphakic Contact lens
  INTERVENTION: aphakic contact lens
- Aphakic Intraocular Lens: optical correction of infant aphakia with aphakic Intraocular Lens
  INTERVENTION: aphakic intraocular lens
Period: Phase 1 (to Age 1 Year)
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Started | 57 | 57
Complete First Endpoint at 1 Year | 57 | 57
Completed | 57 (Age 1 data collection visit) | 57 (Age 1 data collection visit)
Not Completed | 0 | 0
Period: Phase 2 (Age 1 Year to Age 5 Years)
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Started | 57 (Visual acuity assessment at Age 4.5 Years and final visit at Age 5 Years.) | 57 (Visual acuity assessment at Age 4.5 Years and final visit at Age 5 Years.)
Completed | 57 | 56 (Patient lost to follow-up.)
Not Completed | 0 | 1
Period: Phase 3 (Age 10 Years)
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Started | 57 | 56
Completed | 55 | 55
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: months]
  mean/sd | 2.4 (1.6) | 2.5 (1.6) | 2.5 (1.6)
Age, Customized [Number; unit: participants]
  28 - 48 days | 25 | 25 | 50
  49 days - 3.0 months | 17 | 15 | 32
  3.1 - 5.0 months | 9 | 10 | 19
  5.1 - 6.8 months | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 25 | 29 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 48 | 47 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 49 | 48 | 97
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 57 | 57 | 114
Private Insurance [Number; unit: participants]
  No | 20 | 24 | 44
  Yes | 37 | 33 | 70
Qualified for Medicaid [Number; unit: participants]
  No | 40 | 35 | 75
  Yes | 17 | 22 | 39
Pupil Diameter - Cataractous Eye [Mean (Standard Deviation); unit: mm] | 3.3 (1.0) | 3.2 (1.0) | 3.3 (1.0)
Pupil Diameter - Fellow Eye [Mean (Standard Deviation); unit: mm] | 3.5 (0.9) | 3.4 (0.9) | 3.4 (0.9)
Corneal Diameter - Cataractous Eye [Mean (Standard Deviation); unit: mm] | 10.5 (0.7) | 10.5 (0.8) | 10.5 (0.7)
Corneal Diameter - Fellow Eye [Mean (Standard Deviation); unit: mm] | 10.8 (0.6) | 10.8 (0.7) | 10.8 (0.6)
Intraocular Pressure - Cataractous Eye [Mean (Standard Deviation); unit: mmHg] | 12.7 (4.9) | 11.8 (4.9) | 12.2 (4.9)
Intraocular Pressure - Fellow Eye [Mean (Standard Deviation); unit: mmHg] | 12.8 (5.1) | 12.9 (4.3) | 12.9 (4.7)
Keratometric Power - Cataractous Eye [Mean (Standard Deviation); unit: diopters] | 46.4 (2.7) | 46.4 (2.7) | 46.4 (2.7)
Keratometric Power - Fellow Eye [Mean (Standard Deviation); unit: diopters] | 45.5 (1.8) | 45.4 (1.9) | 45.5 (1.8)
Axial Length - Cataractous Eye [Mean (Standard Deviation); unit: mm] | 18.0 (1.3) | 18.1 (1.3) | 18.0 (1.3)
Axial Length - Fellow Eye [Mean (Standard Deviation); unit: mm] | 18.4 (0.9) | 18.7 (0.9) | 18.6 (0.9)
Refractive Error - Fellow Eye [Mean (Standard Deviation); unit: diopters] — Spherical equivalent of the refraction measured under cycloplegia
  diopters | 2.4 (1.8) | 2.3 (2.2) | 2.3 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity was measured by standard objective testing procedures at 12 months of age. Monocular grating acuity was assessed by the traveling examiner with the Teller Acuity Cards. This test uses cards with black-on-white lines of varying widths and a set distance apart in a square with fixed dimensions, so the thinner the lines, the more there will be on any given card (cycles/cm). The ability to see thinner lines indicates better vision. The cards with lines are presented simultaneously with a gray card and the child's visual attention is noted. It is presumed that the child will preferentially look at the card with the stripes as it is more interesting. When the lines are too thin and close together so as to be indistinguishable from the gray card, no preferential looking will be noted. The card with the thinnest lines that the child will look at is recorded as the best visual acuity in logMAR units.
Time Frame: Phase 1 - Age 12 months
Population: The number of participants was determined by the sample size estimate necessary to detect a 0.2 logMAR difference (2 lines on the Snellen chart) in the visual acuity between the two groups.
Measure: Median (Inter-Quartile Range); unit: logMAR units
Groups:
- Aphakic Contact Lens: optical correction of infant aphakia with aphakic Contact lens
  INTERVENTION: use of an external contact lens (CL) to correct the large hyperopic refractive error produced by surgically extracting the natural cataractous lens. As the eye grows, the refractive error changes and the power of the CL can be changed accordingly.
- Aphakic Intraocular Lens: optical correction of infant aphakia with aphakic Intraocular Lens
  INTERVENTION: The refractive error induced by surgical removal of the cataractous natural lens is partially corrected by the implantation of an intraocular lens (IOL) at the time of surgery. This is deemed a permanent correction as the IOL may only be removed in a subsequent surgery.
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 57 | 57
logMAR units | 0.80 [0.66 to 0.97] | 0.97 [0.80 to 1.10]
Statistical Analysis 1: Comparison: Aphakic Contact Lens vs Aphakic Intraocular Lens; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Visual Acuity - Subjective Assessment at Age 4.5 Years.
Description: Visual acuity estimates were standardized by using the Electronic Visual Acuity Tester (EVAT) at each clinical site. The IATS patients were tested at 4.5 years of age allowing the use of the HOTV recognition acuity test. The Amblyopia Treatment Study protocol for presentation and determination of best corrected visual acuity was followed. Monocular visual acuity was evaluated using single letter optotypes with surround bars presented on the EVAT. The staircase procedure of the ATS projects was followed as this has documented success and reliability with this age group. In order to familiarize the subjects with the HOTV matching test, this test was introduced at the 4.0 year visit and the 4.25 year visit by experienced site personnel.
Time Frame: Phase 2 - Age 4.5 Years
Population: One patient in the intraocular lens group was lost to follow-up.at age 18 months. A second patient in that group had developmental delay and the visual acuity could not be assessed. Therefore, the visual acuity measurements at 4.5 years of age are reported for 55 of the 57 patients randomized to the intraocular lens group.
Measure: Median (Inter-Quartile Range); unit: logMAR units
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 57 | 55
logMAR units | 0.90 [0.30 to 1.60] | 0.90 [0.40 to 1.73]
Statistical Analysis 1: Comparison: Aphakic Contact Lens vs Aphakic Intraocular Lens; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Visual Acuity - Subjective Assessment at Age 10 Years.
Description: Visual acuity estimates were standardized by using the Electronic Visual Acuity Tester (EVAT) at each clinical site. The IATS patients were tested at 10.5 years of age allowing the use of the electronic early treatment diabetic retinopathy study (E-ETDRS) testing protocol. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision).
Time Frame: Phase 3 - Age 10.5 Years
Population: Participants who completed the third phase of the study are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: logMAR units
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 55 | 55
logMAR units | 0.86 [0.30 to 1.46] | 0.89 [0.33 to 1.43]
Statistical Analysis 1: Comparison: Aphakic Contact Lens vs Aphakic Intraocular Lens; Test type: Other; p = 0.82, Chi-squared

4. Secondary Outcome: Percent of Patients With 1 or More Intraoperative Complications at Cataract Surgery
Description: Percent of Patients with 1 or More Intraoperative Complications at Cataract Surgery
Time Frame: Cataract surgery immediately after enrollment
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Aphakic Contact Lens: optical correction of infant aphakia with aphakic Contact lens
  INTERVENTION: use of an external contact lens (CL) to correct the large hyperopic refractive error produced by surgically extracting the natural cataractous lens. As the eye grows, the refractive error changes and the power of the CL can be changed accordingly.
  hyperopic correction of infant surgical aphakia with Contact Lens: optical correction of infant surgical aphakia with Contact lens
- Aphakic Intraocular Lens: optical correction of infant aphakia with aphakic Intraocular Lens
  INTERVENTION: At the time of surgery to remove the cataractous natural lens, an intraocular lens was implanted to correct the large hyperopic refractive error induced by the cataract surgery.
  primary implantation of aphakic intraocular lens: optical correction of surgical aphakia with intraocular lens
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 57 | 57
percentage of patients | 11 [4 to 22] | 28 [17 to 42]
Statistical Analysis 1: Comparison: Aphakic Contact Lens vs Aphakic Intraocular Lens; Test type: Superiority; p = 0.03, Fisher Exact

5. Secondary Outcome: Percent of Patients With 1 or More Adverse Events
Time Frame: Study enrollment to age 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 57 | 57
percentage of patients | 56 [42 to 69] | 81 [68 to 90]
Statistical Analysis 1: Comparison: Aphakic Contact Lens vs Aphakic Intraocular Lens; Test type: Superiority; p = 0.008, Fisher Exact

6. Secondary Outcome: Parenting Stress
Description: The PSI is a 120-item validated self-report measure of parenting stress. PSI is a continuous scale measuring stress with a range of 131 (low stress) to 320 (high stress); the average person's stress scores are between 188 and 252.
Time Frame: Phase 1 - 3 months post surgery
Population: All those who completed the PSI 3 months after surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 55 | 53
units on a scale | 197.4 (35.7) | 231.1 (36.8)
Statistical Analysis 1: Comparison: Aphakic Contact Lens vs Aphakic Intraocular Lens; ITT analyses comparing parents of children randomized to receive an IOL to those left aphakic; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 15.7

7. Secondary Outcome: Adherence to Occlusion Therapy
Description: Parental report of the number of hours children wore an patch to occlude the fellow eye.
Time Frame: Phase 1 - 12 months follow-up
Population: Analysis is limited to those with at least 3 reports of adherence before 12 months of age.
Measure: Mean (Standard Deviation); unit: Hours patched per day
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 53 | 53
Hours patched per day | 3.92 (1.55) | 3.63 (1.68)

8. Secondary Outcome: Parenting Stress
Description: as for outcome 6
Time Frame: Phase 1 - Age 12 Months
Population: All those who completed the PSI 3 months after surgery and the PSI at age 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
Number analyzed (Participants) | 43 | 38
units on a scale | 202.6 (34.4) | 208.3 (30.8)
Statistical Analysis 1: Comparison: Aphakic Contact Lens vs Aphakic Intraocular Lens; ITT comparison of mean PSI scores; Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 7.295

ADVERSE EVENTS:
Time Frame: Ocular adverse events occurring the day after enrollment until the follow-up visit at 10.5 years of age are reported.
Arm/Group | Aphakic Contact Lens | Aphakic Intraocular Lens
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 32/57 | 46/57
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aphakic Contact Lens (N=57) | Aphakic Intraocular Lens (N=57)
Lens reproliferation into visual axis (Eye disorders) | 2 (2) | 23 (23)
Pupillary membrane (Eye disorders) | 2 (2) | 16 (16)
Corectopia (Eye disorders) | 1 (1) | 16 (16)
Glaucoma (Eye disorders) | 9 (9) | 11 (11)
Glaucoma suspect (Eye disorders) | 11 (11) | 5 (5)
Contact lens related adverse event (Eye disorders) | 10 (10) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 2 (2) | 5 (5)
Retinal hemorrhage (Eye disorders) | 2 (2) | 3 (3)
Hyphema (Eye disorders) | 1 (1) | 4 (4)
Retained cortex (Eye disorders) | 2 (2) | 3 (3)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Phthisis bulbi (Eye disorders) | 1 (1) | 0 (0)
Corneal edema lasting more than 30 days (Eye disorders) | 0 (0) | 1 (1)
Wound leak or dehisence (Eye disorders) | 0 (0) | 1 (1)
Intraocular lens capture (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT00212134/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT00212134/ICF_001.pdf